CLINICAL TRIAL: NCT04152265
Title: Mycotoxin Exposure and Dietary Habits in Colorectal Cancer Prevention and Development Among Polish Population
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Warmia and Mazury in Olsztyn (Other)
Collaborators: Provincial Specialist Hospital in Olsztyn (Unknown); Ministry of Health Republic of Poland (Unknown)
Responsible Party: Principal Investigator, Tomasz Sawicki, Principal Investigator, University of Warmia and Mazury in Olsztyn
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 6/2019
Record Dates: First submitted 2019-10-28; First posted 2019-11-05 (Actual); Last update posted 2019-11-05 (Actual); Status verified 2019-11

CONDITIONS: Colorectal Cancer, Somatic (Diagnosis)
Keywords: colorectal cancer; zearalenone; mycotoxin; gastrointestinal bacterial
MeSH Terms: conditions — Colorectal Neoplasms; Disease | interventions — Colonoscopy; Surveys and Questionnaires

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No Intervention: Current screening practice. (Other): Patients will be asked to complete the Food Frequency Questionnaire (FFQ) and the questionnaire about The World Health Organization Quality Of Life (WHOQOL-BREF), also and will be collected the demographic and anthropometric data
  Interventions: Other: questionnaires; Other: demographic data collections; Other: anthropometric data collections
- Experimental: Sequential screening strategy (Experimental): People aged between 50-65, will take part in the study. Patients, which will take in a screening colonoscopy, will be divided into two groups according to the result obtained. The first group, will be constitute the patients with a positive test result, while the second group (control) will be constitute the patients with the negative test result. In addition, from the Subjects the samples of blood and faeces will be collected.
  Interventions: Procedure: colonoscopy; Procedure: Collecte the biological samples

INTERVENTIONS:
Procedure: colonoscopy — colonoscopy
  Arms: Experimental: Sequential screening strategy
Other: questionnaires — complete the two questionnaires (Food Frequency Questionnaire (FFQ) and the questionnaire of The World Health Organization Quality of Life (WHOQOL-BREF)
  Arms: No Intervention: Current screening practice.
Other: demographic data collections — completing the demographic questionnaire
  Arms: No Intervention: Current screening practice.
Other: anthropometric data collections — For the determination of anthropometric data will be used a professional body mass composition analyser (Seca,Hamburg, Germany)
  Arms: No Intervention: Current screening practice.
Procedure: Collecte the biological samples — blood and faeces collections
  Arms: Experimental: Sequential screening strategy

SUMMARY:
The aim of the study is the determination of the zearalenone and its metabolites (α and β) level in the blood plasma and faeces of patients at increased risk of cancer, in relation to the nutrition data (FFQ) and information on the quality of life dependent on health (WHOQOL-BREF).

The study is performer within the framework of the Polish Colonoscopy Screening Program. Within the study 100 volunteers between 50 and 65 years of age. while, the colonoscopies will be performed in Provincial Specialist Hospital in Olsztyn. Patients with positive test result, who have been diagnosed with polyps or cancer, will be assigned to risk group. The study has been approved by a local bioethics committee.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged from 50 to 65 years residing in Poland.

Exclusion Criteria:

* subjects requiring long-term care due to somatic, mental retardation or other mental illness.
* history of colorectal resection.

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-11-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Completion of the assigned screening strategy | Within 8 weeks of enrollment
  Completion of the assigned screening strategy within 8 weeks of enrollment defined as:
  * current screening strategy: documented screening colonoscopy.

SECONDARY OUTCOMES:
Analysis of the concentration of the mycotoxin | 5 month
  Determination of the concentration and a profile of the mycotoxin using the high-performance liquid chromatography coupled with the mass spectrometry (HPLC-MS)
Characteristics of gut bacterial | 6 month
  The presence of bacterial DNA in the samples will be confirmed using real-time polymerase chain reaction (RT-PCR). Microbial diversity will be study by sequencing the amplified V3-V4 region of the 16S rRNA gene by using primers 16S. Next, the amplicon pools will be prepared for sequencing and the size and quantity of the amplicon library will be assessed on NGS MiSeq.
Determination of anthropometric data | 4 weeks
  The anthropometric data will be determined using the professional body mass composition analyser. Based on the obtained data will be calculated Body Mass Index (BMI), which will be expressed in kg/m^2

CONTACTS AND LOCATIONS:
Overall Officials: Tomasz Sawicki, PhD, Principal Investigator — Department of Human Nutrition, Faculty of Food Science, University of Warmia and Mazury
Locations (1):
- Provincial Specialist Hospital in Olsztyn, Olsztyn, Poland